CLINICAL TRIAL: NCT04614402
Title: Transcatheter Repair of Tricuspid Regurgitation With Edwards PASCAL Transcatheter Valve Repair System: A European Prospective, Multicenter Post-Market Clinical Follow up
Brief Title: Transcatheter Repair of Tricuspid Regurgitation With Edwards PASCAL Transcatheter Valve Repair System
Acronym: TriCLASP
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-11
Record Dates: First submitted 2020-09-25; First posted 2020-11-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Edwards PASCAL Transcatheter Valve Repair System — The Edwards PASCAL Valve Repair System is indicated for the percutaneous reconstruction of an insufficient tricuspid valve.
Device: Edwards PASCAL Precision Transcatheter Valve Repair System — The Edwards PASCAL Precision Valve Repair System is indicated for the percutaneous reconstruction of an insufficient tricuspid valve.

SUMMARY:
This is a postmarket clinical follow up study on the safety and effectiveness of the Edwards PASCAL Transcatheter Valve Repair System and the Edwards PASCAL Precision Transcatheter Valve Repair System in transcatheter tricuspid valve repair.

DETAILED DESCRIPTION:
The objectives of this clinical study are to collect data on the safety and effectiveness of the PASCAL System and PASCAL Precision System in improving TR, functional status, and quality of life in a post-market setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a candidate for transcatheter tricuspid valve repair as determined by a Heart Team
2. TR grade ≥3+ (5 grade classification)
3. Patient is eligible to receive the PASCAL device per the current approved indications for use

Exclusion Criteria:

1. Tricuspid valve anatomic contraindications, including previous tricuspid valve replacement
2. Severe aortic, mitral, and/or pulmonic valve stenosis and/or regurgitation
3. Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator
4. Any patient considered to be part of a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at or over the age of 18 determined to require percutaneous reconstruction of an insufficient tricuspid valve (TR ≥ 3+) by a Heart Team who assesses patient risk and anatomic suitability for the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major adverse events (MAE rates) | 30 days
  The primary safety endpoint is the proportion of patients with major adverse events (MAEs) at 30 days
Change in tricuspid regurgitation severity (scale of 0-5) by echocardiography | Discharge: defined as discharge or 7 days post-procedure, whichever comes first
  Reduction in TR severity as assessed by TEE pre and post-implant in the procedure room. TR severity compared to baseline will be assessed by TR grade at each follow-up interval.

SECONDARY OUTCOMES:
Volume overload assessed by serial measurements | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  Patient edema questionnaire
Volume overload assessed by serial measurements | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  Body weight in kilogram
Volume overload assessed by serial measurements | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  Edema Assessment (scale 1+ - 4+) grade correspond to mm
Volume overload assessed by serial measurements | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  Ankle circumference measurement in cm
Functional class, functional status, and Quality of life as assessed | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  NYHA classification (I-IV) grade
Functional class, functional status, and Quality of life as assessed | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  6-Minute Walk Test in meter
Functional class, functional status, and Quality of life as assessed | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  5 Level EQ 5D Questionnaire
Functional class, functional status, and Quality of life as assessed | baseline, 30 days, 6 months, 12 months, annually up to 5 years
  Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Baldus, Prof. Dr., Principal Investigator — Herzzentrum Uniklinik Köln, Klinik III für lnnere Medizin
Locations (15):
- Germany (12):
  - Universitätsklinikum Tübingen Innere Medizin III - Kardiologie und Angiologie, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm Innere Medizin II, Ulm, Baden-Wurttemberg
  - Medizinische Klinik I- Campus Grosshadern, München, Bavaria
  - Herzzentrum Universitätsklinikum Köln, Cologne, DEU
  - Westdeutsches Herz- und Gefäßzentrum Klinik für Kardiologie und Angiologie, Essen, Nordrhine Westfalia
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum der Universitätsklinik Bonn, Bonn, North Rhine-Westphalia
  - Heart Centre of the University Leipzig, Leipzig, Saxony
  - Zentralklinik Bad Berka GmbH, Bad Berka, Thuringia
  - UKE Hamburg, Hamburg
  - Kath. Marienkrankenhaus Hamburg gGmbH, Hamburg
  - University Heart Center Lübeck, Lübeck
- Hygeia Hospital, Athens, Greece
- Ospedale del Cuore "G. Pasquinucci", Massa, Italy
- Inselspital, Bern, Switzerland